CLINICAL TRIAL: NCT07365163
Title: Comparative Effects of Deep Breathing Exercises and Volume-oriented Incentive Spirometry on Dyspnea, Functional Endurance, and Pulmonary Function During the Third Trimester of Pregnancy
Brief Title: Breathing Exercises Versus Incentive Spirometry in Third-Trimester Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: University of Lahore Hospital (ULH) (Network)
Responsible Party: Principal Investigator, Adnan Hashim, Doctor of Physical Therapy Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRI/IREB/26/01/0023
Record Dates: First submitted 2026-01-04; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dyspnea During Pregnancy; Physiological Changes in Pregnancy; Reduced Functional Endurance
Keywords: Physical Therapy; Deep Breathing Exercises; Incentive Spirometry; Pregnancy; Third Trimester; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel intervention groups: a deep breathing exercise group or a volume-oriented incentive spirometry group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation to reduce assessment bias. Participants and care providers were not blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Breathing Exercise Group (Experimental): Participants assigned to this arm performed a structured deep breathing exercise program consisting of slow, controlled inhalation and exhalation techniques under supervision during the intervention period.
  Interventions: Other: Deep Breathing Exercises
- Incentive Spirometry Group (Experimental): Participants assigned to this arm performed volume-oriented incentive spirometry exercises using a standard incentive spirometer according to a predefined protocol during the intervention period.
  Interventions: Device: Volume-Oriented Incentive Spirometry

INTERVENTIONS:
Other: Deep Breathing Exercises — Deep breathing exercises focused on diaphragmatic breathing with slow, deep inhalation followed by controlled exhalation. The exercises were performed according to a standardized protocol under supervision.
  Arms: Deep Breathing Exercise Group
Device: Volume-Oriented Incentive Spirometry — Volume-oriented incentive spirometry involved slow, sustained maximal inspiration using an incentive spirometer device to encourage lung expansion and improve respiratory function, performed under supervision according to protocol.
  Arms: Incentive Spirometry Group

SUMMARY:
Shortness of breath (dyspnea) is commonly experienced during the third trimester of pregnancy due to physiological changes affecting the respiratory system. Non-pharmacological breathing interventions are often recommended to improve breathing comfort and functional capacity in pregnant women.

This randomized controlled trial compared the effects of deep breathing exercises and volume-oriented incentive spirometry on dyspnea, functional endurance, and pulmonary function in women during the third trimester of pregnancy. Eligible participants were randomly assigned to one of two intervention groups. One group performed supervised deep breathing exercises, while the other group performed volume-oriented incentive spirometry exercises.

Outcomes were measured before and after the intervention period and included the severity of dyspnea, functional endurance, and pulmonary function parameters. The results of this study aim to provide evidence regarding the effectiveness of simple, safe, and non-invasive breathing interventions for improving respiratory outcomes during late pregnancy.

DETAILED DESCRIPTION:
This study was a randomized controlled trial designed to evaluate and compare the effects of two non-pharmacological respiratory interventions in women during the third trimester of pregnancy. Physiological changes during pregnancy, such as diaphragmatic elevation and increased oxygen demand, can contribute to dyspnea and reduced functional endurance. Safe and effective breathing interventions may help alleviate these symptoms without pharmacological risk.

Eligible pregnant women in their third trimester who met the inclusion criteria were recruited and randomly allocated into two intervention groups using a randomization method. Participants in Group A received a structured deep breathing exercise program, which focused on slow, controlled inhalation and exhalation techniques performed under supervision. Participants in Group B received volume-oriented incentive spirometry training, which encouraged sustained maximal inspiration using a standard incentive spirometer device.

Both interventions were administered according to a predefined protocol over the study period. Outcome measures were assessed at baseline and after completion of the intervention period. Primary outcomes included the assessment of dyspnea severity. Secondary outcomes included measures of functional endurance and pulmonary function.

The study was conducted in accordance with ethical standards and received approval from the institutional ethics review committee. All participants provided informed consent prior to participation. The findings of this study are intended to contribute to evidence-based physical therapy practice by identifying effective, low-risk breathing interventions for managing dyspnea and improving respiratory function during the third trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* - Participants aged between 18 and 40 years
* Blood pressure below 140/90 mmHg
* Not pregnant
* Primigravida women
* Participants in the third trimester of pregnancy
* Able to understand and follow instructions
* Willing to participate and provide informed consent

Exclusion Criteria:

* - History of cardiovascular disorders
* History of respiratory disorders
* History of psychological disorders
* History of medical or surgical conditions involving the nose, throat, diaphragm, or lungs
* Any condition that could interfere with participation in breathing exercises or spirometry

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Functional Endurance | Baseline and at the end of the intervention period (approximately 6 weeks)
  Functional endurance was assessed using the 6-Minute Walk Test (6MWT), which measures the total distance walked by a participant on a flat surface over six minutes. The outcome is reported in meters, with higher values indicating better functional endurance. The minimum possible value is 0 meters, and there is no predefined maximum value.

SECONDARY OUTCOMES:
Forced Expiratory Volume in One Second (FEV₁) | Baseline and at the end of the intervention period (approximately 6 weeks)
  Pulmonary function was assessed using spirometry by measuring Forced Expiratory Volume in one second (FEV₁). FEV₁ is reported in liters, with higher values indicating better pulmonary function.
Forced Vital Capacity (FVC) | Baseline and at the end of the intervention period (approximately 6 weeks)
  Pulmonary function was assessed using spirometry by measuring Forced Vital Capacity (FVC). FVC is reported in liters, with higher values indicating better pulmonary function.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study was conducted as a university-based academic research project with data collected for thesis purposes. The informed consent obtained from participants did not include provisions for public data sharing, and the dataset contains sensitive personal health information. Data will be stored securely at the institution and used only for academic and research purposes in accordance with institutional ethics approval.

REFERENCES:
- [Background] ZAHRA, M. S., SHIMAA, T. T., YOUSSEF, M. S., & EMAD, M. T. (2021). Effect of Deep Breathing on Functional Capacity among Healthcare Workers Wearing FFP2/N95 Filtering Facepiece Respirators. The Medical Journal of Cairo University, 89(September), 1699-1706.
- [Background] Yüksel, F., Guzel, N. A., Taspinar, B., & Balaban, A. (2020). Relationship between trunk muscle endurance, pulmonary function, and respiratory muscle strength in healthy individuals. Türk Fizyoterapi ve Rehabilitasyon Dergisi, 31(3), 255-262.
- [Background] Villarta Jr, R. L., & Asaad, A. S. (2014). Sample Size Determination in an Epidemiologic Study using the EpiTools Web-Based Calculator. Acta Medica Philippina, 48(1).
- [Background] Siraj, S., Israr, S., Jamshed, K., & Tahir, L. (2022). Incidence and Causes of Dyspnea in Pregnant Women: Experience from a Tertiary Care Hospital. Pakistan Journal of Chest Medicine, 28(4), 420-425.
- [Background] Shetty N, Samuel SR, Alaparthi GK, Amaravadi SK, Joshua AM, Pai S. Comparison of Diaphragmatic Breathing Exercises, Volume, and Flow-Oriented Incentive Spirometry on Respiratory Function in Stroke Subjects: A Non-randomized Study. Ann Neurosci. 2020 Jul;27(3-4):232-241. doi: 10.1177/0972753121990193. Epub 2021 Mar 17. PMID 34556964
- [Background] Sewa, D. W., & Ong, T. H. (2014). Pulmonary function test: spirometry. Proceedings of Singapore Healthcare, 23(1), 57-64.
- [Background] Rufaida, Z., Istiqomah, R., & Lestari, S. W. P. (2023). EFFECT OF DEEP BREATH RELAXATION ON THE ANXIETY AMONG THIRD TRIMESTER PREGNANT WOMEN IN MOJOKERTO DISTRICT, INDONESIA: A QUASI EXPERIMENT. Journal of Community Mental Health and Public Policy, 6(1), 41-47.
- [Background] Rafea, A., Wagih, K., Amin, H., El-Sabagh, R., & Yousef, S. (2009). Flow-oriented incentive spirometer versus volume-oriented spirometer training on pulmonary ventilation after upper abdominal surgery. Egyptian Journal of Bronchology, 3(2), 110-118.
- [Background] Pellegrim, C. (2022). Dyspnea, Level of Physical Activity and Social and Emotional Factors in Pregnant Women in the Context of the COVID-19 Pandemic in Portugal Universidade de Aveiro (Portugal)].
- [Background] Moore, Y., Shotton, E., Brown, R., Gremmel, J., Lindsey, S., & Pankey, J. (2018). Effects of incentive spirometry on perceived dyspnea in patients hospitalized with pneumonia. MedSurg Nursing, 27(1), 19-37.
- [Background] Kumar AS, Alaparthi GK, Augustine AJ, Pazhyaottayil ZC, Ramakrishna A, Krishnakumar SK. Comparison of Flow and Volume Incentive Spirometry on Pulmonary Function and Exercise Tolerance in Open Abdominal Surgery: A Randomized Clinical Trial. J Clin Diagn Res. 2016 Jan;10(1):KC01-6. doi: 10.7860/JCDR/2016/16164.7064. Epub 2016 Jan 1. PMID 26894090
- [Background] Hamilton DM, Haennel RG. Validity and reliability of the 6-minute walk test in a cardiac rehabilitation population. J Cardiopulm Rehabil. 2000 May-Jun;20(3):156-64. doi: 10.1097/00008483-200005000-00003. PMID 10860197
- [Background] Gosselink R. Controlled breathing and dyspnea in patients with chronic obstructive pulmonary disease (COPD). J Rehabil Res Dev. 2003 Sep-Oct;40(5 Suppl 2):25-33. doi: 10.1682/jrrd.2003.10.0025. PMID 15074451
- [Background] Gartner-Schmidt JL, Shembel AC, Zullo TG, Rosen CA. Development and validation of the Dyspnea Index (DI): a severity index for upper airway-related dyspnea. J Voice. 2014 Nov;28(6):775-82. doi: 10.1016/j.jvoice.2013.12.017. Epub 2014 Oct 12. PMID 25311596
- [Background] Felton M, Hundley VA, Grigsby S, McConnell AK. Effects of slow and deep breathing on reducing obstetric intervention in women with pregnancy-induced hypertension: a feasibility study protocol. Hypertens Pregnancy. 2021 Feb;40(1):81-87. doi: 10.1080/10641955.2020.1869250. Epub 2021 Jan 19. PMID 33463384
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Elumalai, S., Suganthirababu, P., & Ramalingam, K. (2024). The Effect of Threshold Inspiratory Muscle Training Device and Incentive Spirometry Device for Dyspnoea among Third-Trimester Antenatal Women. Indian Journal of Physiotherapy & Occupational Therapy, 18.
- [Background] Elsayed, S. H., Basset, W. K. M. A., & Fathy, K. A. (2015). Impact of active cycle of breathing technique on functional capacity in patient with bronchiectasis. International Journal of Therapies and Rehabilitation Research, 4(5), 287.
- [Background] Ejikeme C, Nandakumar V, Gotur D. Respiratory physiological changes in pregnancy. Respir Med. 2025 Sep;246:108245. doi: 10.1016/j.rmed.2025.108245. Epub 2025 Jul 3. PMID 40614834
- [Background] Dumitrascu-Biris D, Nzelu D, Dassios T, Nicolaides K, Kametas NA. Chronic hypertension in pregnancy stratified by first-trimester blood pressure control and adverse perinatal outcomes: A prospective observational study. Acta Obstet Gynecol Scand. 2021 Jul;100(7):1297-1304. doi: 10.1111/aogs.14132. Epub 2021 Mar 17. PMID 33609284
- [Background] Delgado, A., Marinho, G., Melo, R. S., Pinheiro, F., & Lemos, A. (2024). Effectiveness of breathing exercises during first stage of labor: A systematic review and meta-analysis. European Journal of Integrative Medicine, 68, 102370.
- [Background] Chaudhary, S., Chaudhary, N. I., Ghewade, B., & Mahajan, G. (2020). The immediate effects of breathing exercises with acapella and incentive spirometer on preventing early pulmonary complications following cabg-a comparitive study. International Journal of Current Research and Review, 12(17), 51-58.
- [Background] Bordeleau M, Vincenot M, Lefevre S, Duport A, Seggio L, Breton T, Lelard T, Serra E, Roussel N, Neves JFD, Leonard G. Treatments for kinesiophobia in people with chronic pain: A scoping review. Front Behav Neurosci. 2022 Sep 20;16:933483. doi: 10.3389/fnbeh.2022.933483. eCollection 2022. PMID 36204486
- [Background] AMOLA, M., PAWARA, S., & KALRA, S. (2019). Effect of Inspiratory Muscle Training and Diaphragmatic Breathing Exercises on Dyspnea, Pulmonary Functions, Fatigue and Functional Capacity in Pregnancy during Third Trimester. Journal of Clinical & Diagnostic Research, 13(8).
- [Background] Alaparthi GK, Augustine AJ, Anand R, Mahale A. Comparison of Diaphragmatic Breathing Exercise, Volume and Flow Incentive Spirometry, on Diaphragm Excursion and Pulmonary Function in Patients Undergoing Laparoscopic Surgery: A Randomized Controlled Trial. Minim Invasive Surg. 2016;2016:1967532. doi: 10.1155/2016/1967532. Epub 2016 Jul 21. PMID 27525116
- [Background] Agrawal A, Karle E, Patel TP, Wilson G, Hofmann H, Sunna R, Krvavac A. A Pregnant Woman Presenting With Progressively Worsening Dyspnea and Pneumothorax. Chest. 2020 Jun;157(6):e193-e196. doi: 10.1016/j.chest.2019.11.035. PMID 32505325